CLINICAL TRIAL: NCT07093983
Title: Coupling Rehabilitation Versus Constraint Induced Movement Therapy in Post Stroke Patients With Upper Limb Impairment
Brief Title: Comparing Two Therapies to Improve Arm Function After Stroke
Acronym: CR vs CIMT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LARAIB AKBAR
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Stroke
Keywords: CouplingRehabilitation; CIMT; Stroke; impairment
MeSH Terms: conditions — Stroke | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constraint-Induced Movement Therapy (CIMT) Group (Experimental): Participants in this group will receive Constraint-Induced Movement Therapy (CIMT) along with conventional physical therapy. CIMT involves structured, task-specific exercises that focus on improving the use of the affected upper limb by restricting the unaffected arm. Sessions will include activities such as fine motor training, reaching tasks, strengthening exercises, and functional movement tasks. Therapy will be delivered three times per week for 12 weeks.
  Interventions: Other: Constraint-Induced Movement Therapy (CIMT)
- Coupling Rehabilitation Group (Experimental): Participants in this group will receive Coupling Rehabilitation along with conventional physical therapy. Coupling Rehabilitation involves bilateral arm training and task-specific activities that encourage coordinated use of both upper limbs to stimulate recovery in the affected arm. Exercises will include trunk-supported reaching, object manipulation, and simulated daily tasks. Therapy will be provided three times per week for 12 weeks.
  Interventions: Other: Coupling Rehabilitation

INTERVENTIONS:
Other: Constraint-Induced Movement Therapy (CIMT) — Participants in this group will receive modified CIMT in combination with conventional physical therapy. The unaffected arm will be restrained to encourage use of the affected upper limb. Task-specific exercises will include fine motor tasks, strengthening, reaching, and functional movement training. Each session will last approximately 45-60 minutes and will be conducted three times per week for 12 weeks.
  Arms: Constraint-Induced Movement Therapy (CIMT) Group
Other: Coupling Rehabilitation — Participants in this group will receive Coupling Rehabilitation in addition to conventional physical therapy. This method involves bilateral arm training and functional tasks designed to improve coordination between both upper limbs, using the unaffected limb to guide movement in the affected one. Exercises will include trunk-supported reaching, object retrieval, and posture-supported task practice. Sessions will occur three times per week for 12 weeks, each lasting approximately 45-60 minutes.
  Arms: Coupling Rehabilitation Group

SUMMARY:
This clinical trial aims to compare the effects of coupling rehabilitation and constraint-induced movement therapy (CIMT) on improving arm function, hand skills, and daily activity performance in people who have upper limb weakness after a stroke. Participants will be randomly assigned to one of two groups and receive 12 weeks of therapy, including either CIMT or coupling rehabilitation along with conventional physical therapy. The study will evaluate which method is more effective in restoring movement and independence by using standardized assessments before, during, and after the intervention. The findings may help guide future rehabilitation approaches for stroke survivors

DETAILED DESCRIPTION:
This study focuses on improving upper limb recovery in people who have experienced a stroke. Stroke often leads to long-term weakness or difficulty using one arm, which can limit a person's ability to perform everyday tasks such as dressing, eating, or writing. The study explores two promising rehabilitation strategies-Constraint-Induced Movement Therapy (CIMT) and Coupling Rehabilitation-that may help improve arm movement, hand coordination, and independence in daily life.

Participants will take part in therapy sessions over a 12-week period, during which they will engage in structured, goal-oriented exercises tailored to their physical abilities. The research team will monitor changes in motor function and hand dexterity through standard assessments administered at the beginning, mid-point, and end of the study. By comparing outcomes between the two groups, the study seeks to identify which therapy method is more effective in promoting functional recovery after stroke, with the goal of enhancing rehabilitation practices in clinical settings.

ELIGIBILITY:
Inclusion Criteria: •Age 40-65 years old

* Patients suffering from Sub acute stroke
* Motor function score at Fugl-Meyer Assessment between 40-60
* Fine motor assessment at Box and Block Test<20
* ADL's assessment at Motor Activity Log:

Amount of use scale<2.5 Quality of movement scale<3

-

Exclusion Criteria:

* Individuals suffering from unstable angina, symptomatic heart failure, or uncontrolled hypertension
* Physician determined unstable cardiovascular conditions
* The patient has been diagnosed as having organ failure, including the heart, kidneys, and lungs
* Patients with any traumatic musculoskeletal injury to upper limbs
* Individuals who are experiencing cognitive impairment as a result of neurological conditions other than stroke.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-05 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in Upper Limb Motor Function Using the Fugl-Meyer Assessment (FMA) | Baseline, 6 weeks, and 12 weeks after start of intervention
  This outcome assesses changes in motor control and function of the affected upper limb using the Fugl-Meyer Assessment, a validated stroke-specific performance test. Higher scores reflect better motor recovery.
Change in Hand Dexterity Using the Box and Block Test (BBT) | Baseline, 6 weeks, and 12 weeks after start of intervention
  This outcome evaluates fine motor skills and hand coordination by measuring the number of blocks a participant can move from one compartment to another in one minute using the affected hand. Higher scores indicate better hand dexterity.
Change in Performance of Daily Activities Using the Motor Activity Log (MAL) | Baseline, 6 weeks, and 12 weeks after start of intervention
  This outcome assesses real-world use of the affected upper limb in daily activities using the MAL questionnaire. It includes two subscales: Amount of Use (AOU) and Quality of Movement (QOM). Higher scores indicate better function and limb use.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Shabbir, PH.D. PT, Principal Investigator — University of Lahore
Locations (1):
- University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP